CLINICAL TRIAL: NCT00668941
Title: Cyclic Versus Daily Teriparatide on Bone Mass
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helen Hayes Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Health Research, Inc. (Other)
Responsible Party: Principal Investigator, Robert Lindsay, Professor of Clinical Medicine, Helen Hayes Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01 AR056651-01A2, 5RO1 ARO5; R01AR056651-01A2 (NIH)
Record Dates: First submitted 2008-04-27; First posted 2008-04-29 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Osteoporosis
Keywords: Bone Density; Bone Turnover; Histomorphometry
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide; Alendronate; Calcium; Cholecalciferol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): Participants in this group will have been treated with alendronate for at least 1 year prior to study entry. Upon study entry, they will receive a continuous regimen of daily teriparatide (20 mcg subcutaneously) for 48 months, in addition to alendronate. Biopsies will be performed at Week 7 or Month 7.5. The participants will then have the option to be followed while taking alendronate alone for 24-48 months.
  Interventions: Drug: Teriparatide; Drug: Alendronate; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D3
- 2 (Experimental): Participants in this group will have been treated with alendronate for at least 1 year prior to study entry. Upon study entry, they will receive a cyclical regimen of teriparatide, in addition to alendronate. Teriparatide will be administered subcutaneously in 20-mcg doses daily for 3 months. They will receive no teriparatide for the following 3 months, and then teriparatide treatment will continue for the 3 months after that. This schedule will continue for 24 months with an aption to all participants to continue cyclic teriparatide for another 24 months. Biopsies will be performed at Week 7 or Month 7.5.
  Interventions: Drug: Teriparatide; Drug: Alendronate; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D3
- 3 (Active Comparator): Participants in this group will have been treated with alendronate for at least 1 year prior to study entry. Upon study entry, they will continue taking alendronate alone. Biopsies will be performed at Week 7 and then participants in this group will be offered teriparatide as part of Group 2 or 3.
  Interventions: Drug: Alendronate; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D3
- 4 (Experimental): Participants in this group will receive a continuous regimen of teriparatide (20 mcg delivered subcutaneously) daily for 48 months. Biopsies will be performed at Week 7 or Month 7.5. At 24 months the participants will then have the option of taking alendronate and remaining in the study for another 24 months.
  Interventions: Drug: Teriparatide; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D3
- 5 (Experimental): Participants in this group will receive a cyclical regimen of teriparatide. Teriparatide will be administered subcutaneously in 20-mcg doses daily for 3 months. They will receive no teriparatide for the following 3 months, and then teriparatide treatment will continue for the 3 months after that. This schedule will continue for 24 months with an option to all participants to continue cyclic teriparatide for another 24 months. Biopsies will be performed at Week 7 or Month 7.5.
  Interventions: Drug: Teriparatide; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D3
- 6 (Active Comparator): Participants in this group will take only calcium and vitamin D supplements. Biopsies will be performed at Week 7. Participants will then be offered the standard care for osteoporosis or they may enter the study in Group 4 or 5.
  Interventions: Dietary Supplement: Calcium; Dietary Supplement: Vitamin D3

INTERVENTIONS:
Drug: Teriparatide — Teriparatide will be given subcutaneously in 20-mcg doses either continuously or cyclically.
  Arms: 1; 2; 4; 5
Drug: Alendronate — Participants will take 70 mg per week of alendronate for 48 months.
  Arms: 1; 2; 3
Dietary Supplement: Calcium — Calcium supplements will be administered in varied amounts for all participants, but each participant will take enough to bring her total daily calcium intake to 1,200 mg.
Dietary Supplement: Vitamin D3 — Vitamin D3 supplements will be administered in varied amounts for all participants, but each participant will take enough to bring her total daily intake to 1,200 mg.

SUMMARY:
Osteoporosis is a disease that affects millions of individuals in the United States and abroad. It leads to decreased bone mass and causes an increased risk of fracture. This study will compare continuous versus cyclic treatment with teriparatide combined with alendronate, another drug for osteoporosis, or teriparatide alone in women with osteoporosis.

DETAILED DESCRIPTION:
Osteoporosis is a serious bone disease that has become an important public health problem. It causes significant loss of bone mass and increases the risk of both fracture and architectural problems with the skeleton. Until recently, the treatments available for osteoporosis primarily prevented further deterioration of bone by reducing the rate of remodeling within the skeleton. This can reduce the risk of fracture by approximately 50%. Teriparatide is a new type of drug for people with osteoporosis who are at high risk of fracture. Teriparatide stimulates bone remodeling and can correct the underlying architectural and bone mass abnormalities that are characteristic of osteoporosis. This study will compare continuous versus cyclic treatment with teriparatide combined with alendronate, another drug for osteoporosis, or teriparatide alone in women with osteoporosis.

All participants have completed a parent study of two years that included a screening visit with a physical exam, blood draw, x-rays, EKG, and distribution of calcium and vitamin D supplements. Participants will be separated into two groups according to the treatment they have undergone over the year prior to study entry. Participants who have taken alendronate for at least 1 year prior to study entry will be assigned to Protocol 1. Participants who have not previously taken alendronate will be assigned to Protocol 2. Participants in both protocols will be randomly assigned to one of the following three biopsy groups: pre-treatment; early; or late. Participants in the pre-treatment biopsy group will have a bone biopsy before treatment begins. Those participants in the early biopsy group will have a biopsy at Week 7 of treatment, and those in the late group will have a biopsy at Month 7.5 of treatment.

Participants will also be randomly assigned to one of three treatment schedules. Participants in Protocol 1 may be assigned to receive alendronate alone for 24 months; teriparatide daily plus alendronate for 24 months; or teriparatide daily on and off for 3 months at a time plus alendronate for 24 months. Participants in Protocol 2 may be assigned to receive only the supplements they were given during the screening visit; teriparatide daily plus alendronate for 24 months; or teriparatide daily on and off for 3 months at a time for 24 months. Participants will attend assessment visits at Weeks 4 and 7 and Months 3, 5, 6, 7.5, 9, 12, 15, 18, 21, and 24. Visits may include bone turnover measurements, bone mass scans, walking tests, questionnaires, CT scans, and blood draws.

A recently funded extension study will extend the treatment period from 24 to 48 months for all consenting. If the individual was assigned to teriparatide daily (with or without alendronate), they will be given alendronate for the 24 to 48 month time period. If the individual was assigned to cyclic teriparatide, they will continue cyclic therapy foro the 24-48 month period (with or without alendronate).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteoporosis or T score below -2 plus one or more osteoporosis related fractures
* Two measurable vertebrae between L1 and L4
* Willing to undergo a single iliac crest biopsy after administration of 4 tetracycline labels

Exclusion Criteria:

* Secondary causes of osteoporosis or presence of a skeletal disorder other than osteoporosis
* Uses drugs likely to affect skeletal or calcium homeostasis
* Multiple vertebral fractures or severe degenerative changes with fewer than two evaluable vertebrae
* Unwilling to undergo a single iliac crest biopsy
* History of allergy to tetracyclines, exposure to tetracyclines within the last year, or any remote long term use of tetracyclines
* Current use of anti-resorptive medicines (other than alendronate for half the female participants)
* Use of hormone therapy, estrogen therapy, raloxifene, or calcitonin within 6 months before study entry
* Use of any bisphosphonate for more than 3 months within 2 years before study entry (only applies to participants in Groups 4, 5, and 6)
* History of a kidney stone within 5 years before study entry or any history of multiple kidney stones
* Hypercalcemia, hypercalciuria, or elevated parathyroid hormone (reduced 25-hydroxyvitamin D will be corrected prior to admission)
* Esophageal ulceration or stricture or known hypersensitivity to bisphosphonates
* History of external radiation therapy
* Unlikely or unable to complete the study, as determined by the investigators
* Illicit drug use or excessive alcohol consumption

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2005-09; Primary Completion 2016-02 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Bone density | 24 and 48 months

SECONDARY OUTCOMES:
Histomorphometry of iliac crest bone biopsies | Measured at Week 7 and Month 7
HRpQCT (tibia, radius) and QCT (spine and hip)and FEA of these QCT scans | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lindsay, MD, PhD, Principal Investigator — Helen Hayes Hospital
Locations (1):
- Helen Hayes Hospital, West Haverstraw, New York, United States

REFERENCES:
- [Derived] Ganapathy A, Nieves JW, Keaveny TM, Cosman F. Effects of four-year cyclic versus two-year daily teriparatide treatment on volumetric bone density and bone strength in postmenopausal women with osteoporosis. Bone. 2023 Feb;167:116618. doi: 10.1016/j.bone.2022.116618. Epub 2022 Nov 21. PMID 36410666
- [Derived] Cosman F, Nieves JW, Roimisher C, Neubort S, McMahon DJ, Dempster DW, Lindsay R. Administration of teriparatide for four years cyclically compared to two years daily in treatment Naive and alendronate treated women. Bone. 2019 Mar;120:246-253. doi: 10.1016/j.bone.2018.10.020. Epub 2018 Oct 21. PMID 30355512